CLINICAL TRIAL: NCT00444626
Title: A Subject- and Evaluator-Blinded, Randomized, Multi-Center Study to Evaluate the Safety and Effectiveness of Injection With DGE Injectable Gel as Compared to an FDA-Approved Dermal Filler in Subjects Undergoing Cutaneous Correction of Nasolabial Folds
Brief Title: A Study to Compare the Safety and Effectiveness of a Non-FDA Approved Device Dermal Gel Extra (DGE) and an FDA Approved Device for the Correction of Nasolabial Folds (NLFs)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Collaborators: Mentor Worldwide, LLC (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DGE00105
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Results first posted 2015-04-22 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Facial Wrinkles at the Nasolabial Folds
Keywords: nasolabial folds; facial wrinkles
MeSH Terms: interventions — Lidocaine, Prilocaine Drug Combination; Lidocaine; Prilocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DGE (Experimental): Participants received DGE in one nasolabial fold (NLF) of one side of their face (blinded, split-face study design) in the Initial Treatment period. Participants who continued into the Repeat Treatment period were treated with DGE as an open-label treatment.
  Interventions: Device: Dermal Gel Extra (DGE); Drug: EMLA Cream
- Restylane (Active Comparator): Participants received Restylane in one nasolabial fold (NLF) of one side of their face (blinded, split-face study design) in the Initial Treatment period.
  Interventions: Device: Restylane; Drug: EMLA Cream

INTERVENTIONS:
Device: Dermal Gel Extra (DGE) — Dermal Gel Extra (DGE) Injectable Gel contains hyaluronic acid with lidocaine. DGE was administered to nasolabial folds via the intradermal route. The Principal Investigator was instructed to inject a sufficient amount of DGE to ensure full correction of the NLF wrinkles (i.e., to the optimal level of correction achievable). Up to 2 touch-up treatments were allowed in the Initial Treatment period.
  Other Names: PREVELLE Lift; hyaluronic acid and lidocaine
  Arms: DGE
Device: Restylane — Restylane was administered to nasolabial folds via the intradermal route. The Principal Investigator was instructed to inject a sufficient amount of Restylane to ensure full correction of the NLF wrinkles (i.e., to the optimal level of correction achievable). Up to 2 touch-up treatments were allowed in the Initial Treatment period.
  Other Names: dermal filler; hyaluronic acid
  Arms: Restylane
Drug: EMLA Cream — EMLA Cream (Eutectic Mixture of Local Anesthetics) is an FDA-approved topical anesthetic comprised of 2.5% each of lidocaine/prilocaine. EMLA Cream was applied in approximately equal amounts prior to all injections of DGE and Restylane.
  Other Names: lidocaine; prilocaine

SUMMARY:
The purpose of this research study is to evaluate the safety and effectiveness of injection with DGE Injectable Gel (hyaluronic acid with lidocaine manufactured by Genzyme Biosurgery) as compared to injection with Restylane (a Food and Drug Administration (FDA) approved dermal filler) in patients undergoing cutaneous correction of the nasolabial folds (NLFs).

DETAILED DESCRIPTION:
This study included an Initial and a Repeat Treatment period.

The Initial Treatment period was a subject and evaluator-blinded, randomized split face study in which subjects received DGE in one nasolabial fold and Restylane in the other nasolabial fold. Both safety and efficacy were evaluated.

In the Repeat Treatment Period, participants received DGE in both NLFs. Safety was evaluated.

ELIGIBILITY:
Inclusion Criteria (abbreviated list):

* Bilateral nasolabial folds (NLF) with severity score of 3 or 4 on the 6 point scale.

Exclusion Criteria (abbreviated list):

* Pregnant/lactating women.
* Subjects who have an allergy to lidocaine, prilocaine or other amide-type anesthetic.
* Had a chemical peel at the NLF area within 4 weeks prior to study entry. In addition, subjects were restricted from undergoing chemical peels at the NLF area for the duration of the study.
* Had any treatment with Botox® injections in the upper 1/3 of the face within 2 weeks prior to entry into the study, or in the lower 2/3 of the face within 24 weeks prior to entry. In addition, subjects were restricted from receiving Botox injections in the face for the duration of the study.
* Received prior therapy to the face and/or neck (e.g., dermabrasion, face-lift, Thermage®,laser resurfacing, contour threads, non-ablative laser treatments) within 24 weeks prior to study entry. In addition, subjects were restricted from undergoing such therapy for the duration of the study.
* Had previous tissue augmentation at the NLF area within 24 weeks prior to study entry. In addition, subjects were restricted from undergoing tissue augmentation at the NLF area for the duration of the study.
* Had previous treatment at the NLF area with permanent implants (e.g., silicone,Softform®) or long-lasting fillers (e.g., RadiesseTM, Sculptra®, ArteFill® [Artecoll], or Bio-AlcamidTM). In addition, subjects were restricted from undergoing treatment with permanent implants or long-lasting fillers at the NLF area for the duration of the study.
* Had evidence of scar-related disease or delayed healing activity within one year prior to study enrollment. (Note: subjects with scars were eligible for study enrollment, although scars at the intended treatment sites were not treated.)
* Had a history of keloid formation.
* Had a history of hypo- or hyperpigmentation of the skin.
* Had any infection, unhealed wound, or active inflammatory process (e.g., skin eruptions such as cysts, pimples, rashes, or hives) at the injection site(s).
* Immunocompromised/immunosuppressed (e.g., HIV-positive, transplant recipient, or presently receiving chemotherapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2007-05; Primary Completion 2008-02 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (6):
- United States (6):
  - Birmingham, Alabama
  - La Jolla, California
  - Miami Beach, Florida
  - Westwood, New Jersey
  - White Plains, New York
  - Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 166 subjects screened, 26 subjects were never randomized.
Groups:
- Combined Arm: Participants received DGE in one nasolabial fold (NLF) on one side of their face and Restylane in one NLF on the other side of their face (blinded, split-face study design) in the Initial Treatment. For participants who continued into the Repeat Treatment Period, they received DGE in both NLFs as an open-label treatment.
Period: Initial Treatment Period
Arm/Group | Combined Arm
Started | 140
Completed | 128
Not Completed | 12
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 9
Period: Repeat Treatment Period
Arm/Group | Combined Arm
Started | 105 (23 subjects withdrew after completing the Initial Treatment and did not enter the Repeat Treatment)
Completed | 105
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Combined Arms: Participants received DGE in one nasolabial fold (NLF) on one side of their face and Restylane in one NLF on the other side of their face (blinded, split-face study design) in the Initial Treatment. For participants who continued into the Repeat Treatment Period, they received DGE in both NLFs as an open-label treatment.
Arm/Group | Combined Arms
Number analyzed (Participants) | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135
  Male | 5
Race/Ethnicity, Customized [Number; unit: participants] — Multiple responses were possible for race as the screening visit CRF stated "check all that apply".
  participants
    American Indian or Alaskan Native | 9
    Asian | 1
    Black or African American | 24
    Native Hawaiian or Other Pacific Islander | 2
    White | 100
    Other | 5
    Not Available | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Blinded Evaluator's Assessment of Nasolabial Fold (NLF) Wrinkle Severity at Week 24
Description: This was a comparison of the mean change between Baseline and the Week 24 score (baseline minus week 24 scores) in the blinded evaluators' assessments of NLF wrinkle severity. A positive value for the mean change indicates an improvement.
  Genzyme 6-Point Grading Scale (GGS) for NLF was used for the assessment. A GGS score of zero indicates no wrinkles and a score of 5 indicates very deep wrinkles with redundant folds.
Time Frame: Week 24
Population: The Full Analysis Set (FAS) population includes all randomized participants who received both study treatments and had some post-treatment effectiveness data. For the effectiveness analyses based on the FAS population, participants were analyzed as randomized. The FAS population was identical to an intent-to-treat population.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: nasolabial folds
Groups:
- Dermal Gel Extra (DGE): Participants received DGE in one nasolabial fold (NLF) of one side of their face (blinded, split-face study design) in the Initial Treatment period. Participants who continued into the Repeat Treatment Period received DGE in all NLFs as an open-label treatment.
Arm/Group | Dermal Gel Extra (DGE) | Restylane
Number analyzed (Participants) | 129 | 129
Number analyzed (nasolabial folds) | 129 | 129
Units on a scale | 1.8 (1.0) | 1.8 (1.1)

2. Secondary Outcome: Participant's Pain Assessment During the Initial Treatment Measured on a Visual Analog Scale (VAS)
Description: The pain experienced by each participant at the time of injection (time 0) and at 15 and 30 minutes after injection during the initial treatment visit was evaluated. Pain was measured using a VAS of 0 mm (no pain) to 100 mm (extreme pain).
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Dermal Gel Extra (DGE) | Restylane
Number analyzed (Participants) | 129 | 129
Units on a scale
  0 time after injection | 23.2 (20.3) | 48.9 (26.0)
  15 minutes after injection | 6.1 (10.1) | 16.3 (18.0)
  30 minutes after injection | 3.3 (7.0) | 7.9 (13.0)

3. Secondary Outcome: Change From Baseline in the Blinded Evaluator's Assessment of Nasolabial Folds (NLF) Wrinkle Severity at Week 36
Description: Mean change between Baseline and the Week 36 score (Baseline minus week 36 scores) in the blinded evaluators' assessments of NLF wrinkle severity. A positive value for the mean change indicates an improvement.
  Genzyme 6-Point Grading Scale (GGS) for NLF was used for the assessment. A GGS score of zero indicates no wrinkles and a score of 5 indicates very deep wrinkles with redundant folds.
Time Frame: Week 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: nasolabial folds
Arm/Group | Dermal Gel Extra (DGE) | Restylane
Number analyzed (Participants) | 127 | 127
Number analyzed (nasolabial folds) | 127 | 127
Units on a scale | 1.3 (1.2) | 1.3 (1.2)

4. Secondary Outcome: Number of Participants With at Least a 1 Point Improvement From Baseline in the Blinded Evaluator's Assessment of Wrinkle Severity at Week 24
Description: Count of participants with at least a 1-point improvement from Baseline in the Genzyme 6-Point Grading Scale (GGS) at Week 24. A GGS score of zero indicates no wrinkles and a score of 5 indicates very deep wrinkles with redundant folds.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Dermal Gel Extra (DGE) | Restylane
Number analyzed (Participants) | 129 | 129
Participants | 114 | 113

5. Secondary Outcome: Participant Product Preference at Week 24
Description: Participants indicated their product preference at Week 24 after Date of Optimal Correction (DOC).
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Dermal Gel Extra (DGE) | Restylane
Number analyzed (Participants) | 129 | 129
Participants | 56 | 68

6. Secondary Outcome: Participant Product Preference at Week 36
Description: Participants indicated their product preference at Week 36 after Date of Optimal Correction (DOC).
Time Frame: Week 36
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Dermal Gel Extra (DGE) | Restylane
Number analyzed (Participants) | 129 | 129
Participants | 62 | 55

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events During the Initial Treatment Period
Description: Counts of participants with treatment-emergent adverse events (AEs) from the time of injection up to Week 36. AEs are presented regardless of relationship to study device and/or procedure.
  If a participant had more than one occurrence of the same AE, he/she was counted only once. The most severe occurrence of an AE, as well as the most extreme relationship of the AE to the device, was indicated in cases of multiple occurrences of the same AE. For AEs by relationship, procedure-related and device-related AEs are not mutually exclusive and therefore are not additive.
Time Frame: Weeks 1-36
Population: Number of patients randomized to initial treatment phase. Safety Population.
Measure: Number; unit: Participants
Groups:
- Dermal Gel Extra (DGE): Participants received DGE in one nasolabial fold (NLF) of one side of their face (blinded, split-face study design) in the Initial Treatment period. Participants who continued into the Repeat Treatment Period, they received DGE in all NLFs as an open-label treatment.
- Non-NLF: Adverse events that did not occur at the nasolabial folds
Arm/Group | Dermal Gel Extra (DGE) | Restylane | Non-NLF
Number analyzed (Participants) | 140 | 140 | 140
Participants
  Patients with at least one Adverse Event (AE) | 99 | 89 | 28
  AEs by Severity - Mild | 47 | 58 | 13
  AEs by Severity - Moderate | 37 | 24 | 10
  AEs by Severity - Severe | 15 | 7 | 5
  AEs by Relationship - Procedure or Device | 98 | 87 | 5
  AEs by Relationship - Procedure Related | 69 | 61 | 3
  AEs by Relationship - Device Related | 91 | 78 | 2
  AEs by Duration - less than or equal to 7 days | 70 | 67 | 5
  AEs by Duration - more than 7 days | 29 | 22 | 23
  AEs by Treatment - No Treatment | 54 | 57 | 6
  AEs by Treatment - Medication | 13 | 8 | 18
  AEs by Treatment - Non-drug Therapy | 32 | 24 | 3
  AEs by Treatment - Hospitalization | 0 | 0 | 1
  Patients with Baseline AEs | 0 | 0 | 0
  Patients with Serious AEs | 0 | 0 | 1
  Patients with Study Discontinuation due to AEs | 0 | 0 | 1
  Number of Deaths | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events During the Repeat Treatment Period
Description: Count of participants with treatment-emergent adverse events (AEs) from the time of injection for the repeat treatment period up to week 47. AEs are presented regardless of relationship to study device and/or procedure.
  If a participant had more than one occurrence of the same AE, he/she was counted only once. The most severe occurrence of an AE, as well as most extreme relationship of the AE to the device, was indicated in cases of multiple occurrences of the same AE. For AEs by relationship, procedure-related and device-related AEs are not mutually exclusive and therefore are not additive.
Time Frame: weeks 36 up to 47 weeks
Population: Safety Population for repeat treatment.
Measure: Number; unit: Participants
Groups:
- Restylane - Dermal Gel Extra (DGE): Participants received Restylane in one nasolabial fold (NLF) of one side of their face (blinded, split-face study design) in the Initial Treatment period. In the Repeat Treatment Period, participants received DGE on both sides of their face. This represents the experience with DGE for the side of the face that was originally treated with Restylane.
Arm/Group | Dermal Gel Extra (DGE) | Restylane - Dermal Gel Extra (DGE) | Non-NLF
Number analyzed (Participants) | 105 | 105 | 105
Participants
  Patients with at least one Adverse Event (AE) | 55 | 52 | 9
  AEs by Severity - Mild | 32 | 34 | 5
  AEs by Severity - Moderate | 19 | 15 | 2
  AEs by Severity - Severe | 4 | 3 | 2
  AEs by Relationship - Procedure or Device (DGE) | 54 | 50 | 2
  AEs by Relationship - Procedure Related | 50 | 46 | 2
  AEs by Relationship - Device (DGE) Related | 51 | 47 | 2
  AEs by Duration - less than or equal to 7 days | 44 | 44 | 7
  AEs by Duration - more than 7 days | 11 | 8 | 2
  AEs by Treatment - No Treatment | 41 | 40 | 3
  AEs by Treatment - Medication | 7 | 5 | 6
  AEs by Treatment - Non-drug Therapy | 7 | 7 | 0
  AEs by Treatment - Hospitalization | 0 | 0 | 0
  Patients with a Serious AEs | 0 | 0 | 1
  Patients with Study Discontinuation due to AEs | 0 | 0 | 0
  Number of Deaths | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Initial Treatment Period (week 1 to week 36) and Repeat Treatment Period (week 36 up to week 47)
Description: Participant counts of AEs are broken out by Initial Treatment Period and Repeat Treatment Period. Then further summarized as AEs occurring at the nasolabial fold initially treated with DGE, the nasolabial fold initially treated with Restylane, and AEs that did not occur at the nasolabial folds.
Groups:
- Dermal Gel Extra (DGE): Initial Treatment Period: Adverse events that occurred at the nasolabial fold treated with DGE, and occurred during the Initial Treatment Period regardless of relationship to DGE treatment.
- Restylane: Initial Treatment Period: Adverse events that occurred at the nasolabial fold treated with Restylane, and occurred during the Initial Treatment Period regardless of relationship to Restylane treatment.
- Non-NLF: Initial Treatment Period: Adverse events that did not occur at the nasolabial folds, and occurred during the Initial Treatment Period regardless to relationship to either DGE or Restylane treatment.
- Dermal Gel Extra (DGE) - Repeat Treatment Period: Adverse events that occurred at the nasolabial fold that was treated with DGE in the Initial Treatment Period, and occurred during the Repeat Treatment Period regardless of relationship to DGE treatment.
- Restylane - Dermal Gel Extra (DGE) - Repeat Treatment Period: Adverse events that occurred at the nasolabial fold that was treated with Restylane in the Initial Treatment Period, and occurred during the Repeat Treatment Period regardless of relationship to DGE treatment.
- Non-NLF: Repeat Treatment Period: Adverse events that did not occur at the nasolabial folds, and occurred during the Repeat Treatment Period regardless to relationship to DGE treatment.
Arm/Group | Dermal Gel Extra (DGE): Initial Treatment Period | Restylane: Initial Treatment Period | Non-NLF: Initial Treatment Period | Dermal Gel Extra (DGE) - Repeat Treatment Period | Restylane - Dermal Gel Extra (DGE) - Repeat Treatment Period | Non-NLF: Repeat Treatment Period
Serious Adverse Events (participants affected / at risk) | 0/140 | 0/140 | 1/140 | 0/105 | 0/105 | 1/105
Other Adverse Events (participants affected / at risk) | 99/140 | 89/140 | 28/140 | 55/105 | 52/105 | 9/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dermal Gel Extra (DGE): Initial Treatment Period (N=140) | Restylane: Initial Treatment Period (N=140) | Non-NLF: Initial Treatment Period (N=140) | Dermal Gel Extra (DGE) - Repeat Treatment Period (N=105) | Restylane - Dermal Gel Extra (DGE) - Repeat Treatment Period (N=105) | Non-NLF: Repeat Treatment Period (N=105)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 — Reported by investigator as unrelated to study device.
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 — Reported by investigator as unrelated to study device.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dermal Gel Extra (DGE): Initial Treatment Period (N=140) | Restylane: Initial Treatment Period (N=140) | Non-NLF: Initial Treatment Period (N=140) | Dermal Gel Extra (DGE) - Repeat Treatment Period (N=105) | Restylane - Dermal Gel Extra (DGE) - Repeat Treatment Period (N=105) | Non-NLF: Repeat Treatment Period (N=105)
Injection site swelling (General disorders) | 78 | 69 | 0 | 47 | 47 | 0
Injection site pain (General disorders) | 61 | 57 | 0 | 34 | 32 | 0
Injection site bruising (General disorders) | 35 | 29 | 0 | 23 | 23 | 0
Injection site erythema (General disorders) | 30 | 27 | 0 | 33 | 33 | 0
Injection site nodule (General disorders) | 12 | 6 | 0 | 3 | 0 | 0
Injection site pruritus (General disorders) | 11 | 8 | 0 | 6 | 7 | 0
Injection site anaesthesia (General disorders) | 6 | 1 | 0 | 0 | 0 | 0
Injection site induration (General disorders) | 2 | 0 | 0 | 1 | 0 | 0
Injection site paraesthesia (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Injection site discolouration (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Injection site discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Injection site dryness (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 1 | 0 | 0 | 1 | 0 | 0
Injection site inflammation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Injection site papule (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Cyst (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 4 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Injection site pustule (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Open wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Postoperative constipation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Resorption bone increased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 3 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Allergy to arthropod bite (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bone density decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Intraocular pressure increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal investigators (PI) will give Genzyme a draft manuscript or draft publication 60 days before publication. Genzyme will make every reasonable attempt to review publication or manuscript and give feedback in such 60 day period. PI will not use Genzyme confidential information without prior written consent.